CLINICAL TRIAL: NCT05486117
Title: A Phase 1 Clinical Trial to Evaluate the Pharmacokinetics of Twice-daily Applications of Delgocitinib Cream 20 mg/g for 1 Week in Adult Subjects With Moderate to Severe Chronic Hand Eczema.
Brief Title: Pharmacokinetics of Delgocitinib 20 mg/g Cream in Subjects With Chronic Hand Eczema
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LP0133-2285; 2022-000782-40 (EudraCT Number); U1111-1284-2254 (Other: World Health Organization (WHO))
Record Dates: First submitted 2022-07-18; First posted 2022-08-03 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2022-01

CONDITIONS: Chronic Hand Eczema
MeSH Terms: interventions — delgocitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Delgocitinib cream 20 mg/g (Experimental): Twice-daily topical application for 8 days
  Interventions: Drug: Delgocitinib

INTERVENTIONS:
Drug: Delgocitinib — Cream for topical application 20 mg/g

SUMMARY:
The purpose of the trial is to test how much delgocitinib enters the body over a given time period after application of delgocitinib cream in patients with moderate to severe hand eczema.

Delgocitinib is a cream that suppresses specific processes in the body's response to diseases like CHE, such as inflammation. Everyone in the trial will use delgocitinib cream.

The trial will last up to 7 weeks and there will be 6 visits and a phone call. There will be a screening period of up to 4 weeks, a treatment period (with blood sampling) of 11 days and a safety follow-up phone call 11 days after the last visit.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or above at screening.
* Diagnosis of CHE, defined as hand eczema that has persisted for more than 3 months or returned twice or more within the last 12 months.
* Disease severity graded as moderate to severe at screening and baseline according to IGA-CHE (i.e. an IGA-CHE score of 3 or 4).
* Subjects who have a documented recent history of inadequate response to treatment with topical corticosteroids (TCS) (at any time within 1 year before the screening visit) or for whom TCS are documented to be otherwise medically inadvisable (e.g. due to important side effects or safety risks).
* Subjects adherent to standard non-medicated skin care including avoidance of known and relevant irritants and allergens.

Exclusion Criteria:

* Concurrent skin diseases on the hands, e.g. tinea manuum.
* Active atopic dermatitis (AD) requiring medical treatment in regions other than the hands and feet.
* Active psoriasis on any part of the body.
* Hyperkeratotic hand eczema in combination with a history of psoriasis on any part of the body.
* Clinically significant infection (e.g. impetiginised hand eczema) on the hands.
* Systemic treatment with immunosuppressive drugs (e.g. methotrexate, cyclosporine, azathioprine), immunomodulating drugs, retinoids (e.g. alitretinoin), or corticosteroids within 28 days prior to baseline (steroid eyedrops and inhaled or intranasal steroids corresponding to up to 1 mg prednisolone for allergic conjunctivitis, asthma, or rhinitis are allowed).
* Use of tanning beds, phototherapy (e.g. ultraviolet B [UVB], ultraviolet A1 [UVA1], psoralen ultraviolet A [PUVA]), or bleach baths on the hands within 28 days prior to baseline.
* Cutaneously applied treatment with immunomodulators (e.g. phosphodiesterase 4 [PDE-4] inhibitors, pimecrolimus, tacrolimus) or TCS on the hands within 14 days prior to baseline.
* Use of systemic antibiotics or cutaneously applied antibiotics on the hands within 14 days prior to baseline.
* Cutaneously applied treatments in regions other than the hands, which could interfere with clinical trial evaluations or pose a safety concern within 7 days prior to baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2022-11-22 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve 0-12 hours post dose at Day 1 and Day 8 (AUC0-12). | 0-12 hours post dose at Day 1 and Day 8
Maximum observed concentration (Cmax) at Day 1 and at Day 8 (0-12 hours post-dose). | Day 1 and at Day 8 (0-12 hours post-dose)

SECONDARY OUTCOMES:
Time to reach maximum observed concentration (tmax) at Day 1 and Day 8 (0-12 hours post-dose). | Day 1 and Day 8 (0-12 hours post-dose).
Terminal elimination half-life (t1/2) at Day 8. | Day 8.
Number of treatment-emergent adverse events (AEs) from baseline to Day 22 per subject. | Baseline to Day 22

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (1):
- LEO Investigational Site, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thaci D, Gooderham M, Lovato P, Madsen DE, Soehoel A, Bissonnette R. Systemic exposure and bioavailability of delgocitinib cream in adults with moderate to severe Chronic Hand Eczema. J Eur Acad Dermatol Venereol. 2025 Sep;39(9):1612-1621. doi: 10.1111/jdv.20777. Epub 2025 Jun 17. PMID 40525591